CLINICAL TRIAL: NCT00802412
Title: Topiramate to Aid Smoking Cessation in Recovering Alcohol Dependent Men
Brief Title: Topiramate to Aid Smoking Cessation in Alcohol Dependent Men
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEUA-003-08S
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Nicotine Dependence; Alcohol Dependence
Keywords: tobacco use disorders; alcoholism
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Other): The subjects for the proposed study will be 180 currently smoking, treatment-seeking male veterans with alcohol and nicotine dependence. Ninety subjects will be randomized to the topiramate arm and 90 subjects will be randomized to the placebo group.
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): 90 participants, will receive matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — Topiramate will be titrated over 5 weeks to a maximum dosage of 200 mg according to the following schedule: 25mg daily for days 1-7, 50mg daily for days 8-14, 75mg daily for days 15-21, 100mg daily for days 22-28, 150mg daily for days 29-35, 200mg daily for days 36-42. Maximum dosage will be maintained for 6 weeks, followed by a one-week taper-off period (100mg daily for 4 days and 50mg daily for 3 days).
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo — Placebo/study medication will be administered in opaque capsules in an identical fashion to maintain the double-blind study design.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether topiramate is effective as an aid to smoking cessation for recovering alcohol dependent men.

DETAILED DESCRIPTION:
This study is a 12-week, double-blind, placebo-controlled trial to test the efficacy of topiramate versus placebo as an aid to smoking cessation for recovering alcohol dependent men. Another aim of the study is to explore whether or not topiramate reduces relapse to alcohol use in patients with comorbid alcohol and nicotine dependence. All participants will receive a standardized psychosocial intervention in combination with the medication (or placebo). Following completion of the treatment phase of the study, participants will enter a 24-week follow-up period during which the longer-term outcome of the intervention will be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if they:

* are 18-70 years of age, inclusive;
* are male outpatients with a diagnosis of DSM-IV-TR nicotine dependence and alcohol dependence in early full remission (1-36 months abstinence);
* are current tobacco smokers who smoke an average of 10 or more cigarettes per day in the two months prior to the screening visit;
* are motivated to try to quit smoking and maintain abstinence from alcohol and other illicit drugs;

Exclusion Criteria:

Subjects will be excluded if they:

* have any clinically significant laboratory evidence of hematologic, hepatic, cardiovascular, renal, pulmonary, or thyroid disease;
* have a current significant neurologic, hepatic, renal, gastrointestinal, pulmonary, metabolic, cardiovascular, infectious, or endocrine disease;
* have a history of known hypersensitivity to topiramate;
* in the investigator's judgment, pose a current suicidal or homicidal risk;
* have taken any investigational drug within 30 days of baseline; and
* have a current seizure disorder or a history of severe alcohol withdrawal (alcohol withdrawal seizures, hallucinations / illusions, delirium tremens).

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-01; Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Anthenelli, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

REFERENCES:
- [Derived] Anthenelli RM, Heffner JL, Wong E, Tibbs J, Russell K, Isgro M, Dinh E, Wehrle C, Worley MJ, Doran N. A Randomized Trial Evaluating Whether Topiramate Aids Smoking Cessation and Prevents Alcohol Relapse in Recovering Alcohol-Dependent Men. Alcohol Clin Exp Res. 2017 Jan;41(1):197-206. doi: 10.1111/acer.13279. Epub 2016 Dec 28. PMID 28029173
- See also: Click here for more information about this study: Topiramate to Aid Smoking Cessation in Recovering Alcohol Dependent Men — http://www.pac-tarc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topiramate | Placebo
Started | 65 | 67
Completed | 63 | 66
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Topiramate: Received active topiramate
- Placebo: Received placebo
- Total: Total of all reporting groups
Arm/Group | Topiramate | Placebo | Total
Number analyzed (Participants) | 63 | 66 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (9.0) | 46.9 (9.8) | 47.0 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 63 | 66 | 129
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 32 | 40 | 72
Region of Enrollment [Number; unit: participants]
  United States | 63 | 66 | 129
Fagerstrom [Mean (Standard Deviation); unit: units on a scale] — Scores on the Fagerstrom Test for Nicotine Dependence range from 0 to 10, with higher scores indicating greater nicotine dependence.
  units on a scale | 5.4 (2.0) | 6.1 (1.6) | 5.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: 4-week Continuous Abstinence From Smoking
Description: This measure indicates the proportion of participants who did or did not smoke any cigarettes during the final 4 weeks of treatment, which represented weeks 8-12 of study participation.
Time Frame: Weeks 8-12 of treatment.
Measure: Number; unit: percentage of participants abstinent
Groups:
- Topiramate: 12 weeks of topiramate (up to 200 mg/day) plus smoking cessation treatment, with 24-week follow up.
- Placebo: 12 weeks of placebo plus behavioral smoking cessation treatment, with 24 week follow up.
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 63 | 66
percentage of participants abstinent | 7.9 | 10.6

2. Secondary Outcome: Percent Relapsing to Any Drinking or Illicit Drug Use
Description: Alcohol or illicit drug use during treatment or follow up.
Time Frame: 12-week treatment phase, 36-week combined treatment and follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Topiramate | Placebo
Number analyzed (Participants) | 63 | 66
percentage of participants | 31.8 | 27.3
Statistical Analysis 1: Comparison: Topiramate vs Placebo; Test type: Superiority or Other; p = 0.51, Regression, Logistic; Odds Ratio (OR) = 1.60, 95% CI 2-sided [0.4 to 6.5]
Statistical Analysis 2: Comparison: Topiramate vs Placebo; Test type: Superiority or Other; p = .45, Regression, Cox; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.66 to 2.55]

ADVERSE EVENTS:
Arm/Group | Topiramate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 3/66
Other Adverse Events (participants affected / at risk) | 46/63 | 49/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=63) | Placebo (N=66)
alcohol relapse with suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) — 1 participant in the topiramate group experienced an alcohol relapse that included suicidal ideation.
alcohol relapse (Psychiatric disorders) | 0 (0) | 2 (2) — 2 participants in the placebo group experienced relapses to alcohol
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Topiramate (N=63) | Placebo (N=66)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (13)
Headache (General disorders) | 12 (15) | 8 (11)
Paresthesia (Nervous system disorders) | 6 (6) | 12 (12)
Loss of appetite (General disorders) | 9 (9) | 4 (4)
Reduced concentration (Psychiatric disorders) | 8 (8) | 6 (6)
Dysgeusia (General disorders) | 7 (9) | 6 (6)
Dizziness (General disorders) | 4 (4) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 7 (8)
Somnolence (General disorders) | 6 (6) | 5 (5)
Depression (Psychiatric disorders) | 6 (6) | 3 (3)

LIMITATIONS AND CAVEATS:
Dually-dependent male smokers with high rates of SUDs and psychiatric disorders, thus not generalizable to other populations; topiramate dose lower than the dose found to reduce smoking in active alcoholics; attrition may have impacted results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No